CLINICAL TRIAL: NCT07274020
Title: Effectiveness and Safety of Long-Term Intermittent Moxifloxacin Eradication Therapy in Non-Cystic Fibrosis Bronchiectasis: A 12-Month Randomized Controlled Trial
Brief Title: Long-Term Safety and Efficacy of Moxifloxacin in Bronchiectasis Patients
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Montaser Gamal Ahmed, Lecturer of Chest Diseases and Tuberculosis, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASSIUT-CH-MOXI-BE-25
Record Dates: First submitted 2025-10-01; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Bronchiectasis, Non-Cystic Fibrosis
MeSH Terms: conditions — Bronchiectasis | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intermittent Moxifloxacin + Standard Care (Experimental): Participants will receive moxifloxacin 400 mg orally once daily for 7 days every 8 weeks (total 6 cycles over 12 months) in addition to guideline-based standard care
  Interventions: Drug: Intermittent Moxifloxacin + Standard Care
- Standard Care (Control) (Active Comparator): Participants will receive guideline-based standard care without long-term suppressive antibiotics.
  Interventions: Other: Standard Care (in control arm)

INTERVENTIONS:
Drug: Intermittent Moxifloxacin + Standard Care — Moxifloxacin 400 mg orally once daily for 7 days every 8 weeks (total 6 cycles over 12 months), in addition to guideline-based standard care
  Arms: Intermittent Moxifloxacin + Standard Care
Other: Standard Care (in control arm) — Participants will receive guideline-based management of bronchiectasis without long-term suppressive antibiotics.
  Arms: Standard Care (Control)

SUMMARY:
Bronchiectasis is a chronic respiratory disease characterized by recurrent infections, inflammation, and progressive lung damage. Frequent exacerbations are associated with increased morbidity, accelerated lung function decline, and reduced quality of life. Preventing exacerbations is a key therapeutic goal. Moxifloxacin, a fluoroquinolone antibiotic with broad-spectrum activity, may play a role in intermittent eradication therapy to reduce bacterial load, achieve microbiological clearance, and minimize exacerbation frequency.

This randomized controlled trial will evaluate the effectiveness and safety of long-term intermittent moxifloxacin therapy compared with standard care in patients with non-cystic fibrosis bronchiectasis.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age.
* Confirmed diagnosis of non-cystic fibrosis bronchiectasis by high-resolution CT (HRCT).
* History of ≥2 bronchiectasis exacerbations in the previous 12 months.

Exclusion Criteria:

* Diagnosis of cystic fibrosis-related bronchiectasis.
* Known hypersensitivity or contraindication to fluoroquinolones (including moxifloxacin).
* Severe hepatic impairment or severe renal impairment (eGFR <30 mL/min/1.73 m²).
* Pregnancy or breastfeeding.
* History of significant QT prolongation, arrhythmia, or concurrent use of QT-prolonging drugs.
* Use of long-term suppressive antibiotics for bronchiectasis in the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Exacerbation frequency | 12 months
  Number of acute bronchiectasis exacerbations per patient during follow-up

SECONDARY OUTCOMES:
Microbiological clearance | 12 months
  Rate of clearance of Pseudomonas aeruginosa and other pathogens from sputum cultures
Change in FVC | Baseline and 12 months
  Change in Forced vital capacity

CONTACTS AND LOCATIONS:
Overall Officials: montaser gamal ahmed, gamal ahmed, Principal Investigator — Assiut University
Locations (1):
- Assiut University hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No